CLINICAL TRIAL: NCT04247932
Title: Pathways to the Labor Market for Long-term Unemployed: a Comparison of Labor Market Interventions Effects Mechanisms and Implementation
Brief Title: Pathways to Employment for the Long-term Unemployed
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Göteborg University (Other)
Collaborators: Swedish Council for Working Life and Social Research (Other)
Responsible Party: Sponsor
Other Study IDs: 2018-01324
Record Dates: First submitted 2020-01-27; First posted 2020-01-30 (Actual); Last update posted 2020-07-24 (Actual); Status verified 2020-07

CONDITIONS: Unemployment
Keywords: Adolescent; Disabled Persons; Immigrants

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Municipal: Individual participants receiving active labor market intervention from municipal providers
  Interventions: Behavioral: Active labor market intervention
- Non-profit: Individual participants receiving active labor market intervention from non-profit providers
  Interventions: Behavioral: Active labor market intervention
- Register: Matched sample from register data, no intervention provided

INTERVENTIONS:
Behavioral: Active labor market intervention — Behavior change intervention
  Groups: Municipal; Non-profit

SUMMARY:
This project's aims are twofold (1) to uncover and define the underlying theories of change guiding competing active labor market programs (ALMP) in Sweden, and (2) to assess the relative effectiveness of these competing programs in a theory-based non-randomized controlled trial. The purpose is to assess the extent to which competing ALMPs are effective in moving long-term unemployed individuals (i.e. unemployed for 6 months or more) closer to the labor-market.

DETAILED DESCRIPTION:
Long-term unemployment has a profound impact on the health and wellbeing of individuals, families, and communities. In addition, the effects of long-term unemployment have been found to impact subgroups differently. Today there is scant knowledge on the mechanisms that are influential in moving individuals from long-term unemployment closer to the labor market. This study is designed to answer six research questions using a variety of methods (mixed-methods) and outcome measures (self-report, official register). In addition, this study leverages official register data to construct an untreated control group. This study will assess the extent to which an emerging theory of becoming job ready holds under experimental scrutiny.

This project will engage ALMP program administrators and service providers in semi-structured interviews. A total of 6 competing ALMPs will be included in the study. The transcribed interview material will be used as a basis for program theory reconstruction. All specified program theories will be presented back to program stakeholders for validation. ALMP program effectiveness will be assessed quasi-experimentally with pre- (T1) and posttest (T2) collection of self-reported data. Additionally, official register data from the Longitudinal integrated database for health insurance and labor market studies (LISA) will be collected for all participants. In addition, a matched sample will be collected from LISA to be used as a non-treated control group on final policy outcomes (e.g., employment, salary/wage). This study also assesses program implementation and economic outcomes of competing the competing ALMPs.

ELIGIBILITY:
Inclusion Criteria:

* Unemployed for a period of at least 6 months, and
* 25 years old or younger, or
* born outside of Sweden, or
* 55 years old or older without higher education, or
* has a disability (physical, intellectual, neuropsychiatric, or mental) and
* receives social insurance benefits, or
* receives social welfare benefits

Exclusion Criteria:

* referred for services primarily by the Department of Justice

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All individuals receiving intervention from participating service providers during the inclusion period that meet the inclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2020-09-01 (Estimated); Primary Completion 2021-06 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Change in employment and earnings | baseline, 6 months post baseline
  Employment and earnings data collected from official register data

SECONDARY OUTCOMES:
Change in general health | baseline, 6 months post baseline
  Self report on the General Health Questionnaire (GHQ-12)
Change in resilience | baseline, 6 months post baseline
  Self report on the Resilience Scale (RS-14)
Change in perceived employment obstacles | baseline, 6 months post baseline
  Self-report on the Perceived Employment Barriers Scale (PEBS-20)
Change in perceived employment hope | baseline, 6 months post baseline
  Self-report on the Employment Hope Scale (EHS-14)

CONTACTS AND LOCATIONS:
Overall Officials: Mikaela Starke, PhD, Principal Investigator — Department of Social Work, Gothenburg University

IPD SHARING:
Plan to Share IPD: Yes
De-identified participant data for primary and secondary outcome measures will be made available.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data will be made available within 6 months of study completion
Access Criteria: Data access requests will be reviewed and must be accompanied by an ethical approval to use data.